CLINICAL TRIAL: NCT05886868
Title: A Phase I, International, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of BL0020 as A Single Agent in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of BL0020, a Novel Anti-tumor Drug, in Adult Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Best-Link Bioscience, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL0020-101
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BL0020 (Experimental): Dose Escalation Stage: BL0020 will be administered via intravenous infusion on days 1 of a 21-days treatment cycle.
  Dose Expansion Stage: Maximum tolerated dose or the recommended Phase 2 dose (RP2D) from dose escalation Stage.
  Interventions: Drug: BL0020

INTERVENTIONS:
Drug: BL0020 — Dose Escalation Stage: BL0020 will be administered via intravenous infusion on days 1 of a 21-days treatment cycle.
  Dose Expansion Stage: Maximum tolerated dose or the recommended Phase 2 dose (RP2D) from dose escalation Stage.

SUMMARY:
This is the first in human study of BL0020, and the primary objective is to evaluate the safety and tolerability, and determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of BL0020 as a single agent in patients with advanced solid tumors.

This study consists of two parts: Part A (dose escalation stage) and Part B (dose expansion stage).

The study includes screening, treatment and follow-up periods.

In part A, "3+ 3" will be used for dose escalation.

In part B, the dose level and/or enrolled patient population for dose-expansion may be adjusted based on available data on the safety, PK and preliminary efficacy gained from the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study, be able to understand the requirements of a clinical study, and sign informed consent form.
2. Aged ≥ 18 years, male and female.
3. Patients with histologically or cytologically confirmed, unresectable or metastatic advanced solid tumors that have failed despite standard therapy or have no standard therapy exists. TNBC, SCLC, and pancreatic cancer are preferred for the dose expansion phase.
4. Patients with at least one measurable lesion per RECIST (v1.1) (applicable to the Part B: dose-expansion stage only).

   Note: Measurable lesions cannot be selected from the following sites in principle: having received prior radiotherapy or having received other local therapy. If a target lesion at a site that has received prior radiotherapy or other local therapy is the only optional lesion, the progression of the lesion shall be confirmed by the investigator.
5. Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1 at screening.
6. Life expectancy period ≥ 12 weeks.
7. A male patient must agree to use adequate contraception from screening through at least 3 months after the last dose of investigational product BL0020. Male subjects must also agree not to donate sperm from screening through at least 3 months after the dose of investigational product BL0020. Refer to Section 5.5 for more information on highly effective methods of contraception.
8. Women of childbearing potential must have a negative pregnancy test prior to the dosing administration, and agree to use adequate contraception from screening through at least 6 months after the last dose of investigational product BL0020. A female participant of non-childbearing potential will have had at least 12 continuous months of natural (spontaneous) amenorrhoea, follicle stimulating hormone (FSH) level > 40 mIU/mL at screening, and an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms); or have had surgical bilateral oophorectomy, hysterectomy or bilateral tubal ligation beyond 6 weeks prior to screening. Refer to Section 5.5 for more information on highly effective methods of contraception.

Exclusion Criteria:

1. Patients with symptomatic central nervous system (CNS) metastases or carcinomatous meningitis.
2. Patients who have a history of another primary malignancy (with the exception of subjects with cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ of uterine cervix). A patient who has had no evidence of disease from another primary cancer for 3 or more years is allowed to participate in the study.
3. Patients whose pericardial effusion, pleural effusion or ascites remain uncontrollable after intervention.
4. Patients with a history of allogeneic transplantation of organs, bone marrow or stem cell.
5. Patients with Gilbert's syndrome disease.
6. Patients with homozygous for UGT1A1*28 or UGT1A1*6 (only applicable to the patients in 3+3 dose-escalation cohorts at Part A).
7. Patients who have impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   * New York Heart Association class III-IV for cardiac insufficiency or left ventricular ejection fraction < 50% (if the LVEF data is available).
   * Patients with poorly controlled arrhythmia: QTc interval > 480 ms calculated by Fridericia's formula, or congenital syndrome of prolonged QT interval.
   * Any of the following within 6 months prior to the enrollment: myocardial infarction, severe or unstable angina, congestive heart failure, cerebrovascular accident (including transient ischemic attack), symptomatic pulmonary embolism or other clinically significant thromboembolic disease, or coronary artery bypass graft.
   * Clinically significant resting bradycardia.
   * Patients with other clinically significant cardiovascular disease who were assessed as unsuitable for this study by the investigator.
8. Patients with active chronic inflammatory bowel disease at screening (such as Ulcerative Colitis, Crohn's disease), ≥ grade 2 anorexia, nausea, vomiting or signs of intestinal obstruction. Or patients with a history of intestinal obstruction, gastrointestinal perforation, or clinically significant gastrointestinal bleeding within the 6 months prior to enrollment.
9. Known history of clinically significant active Chronic Obstructive Pulmonary Disease (COPD), or other moderate-to-severe chronic respiratory illness present within 6 months.
10. Patients who have a known diagnosis of Human Immunodeficiency Virus (HIV) infection or HIV antibody test positive in screening.
11. Patients with active hepatitis C or chronic hepatitis B at screening ("active hepatitis" defined as HCV RNA level ≥ 200 IU/mL for hepatitis C or HBV DNA level ≥ 2000 IU/mL for hepatitis B at screening). In addition, eligible hepatitis B or hepatitis C patients must agree to antiviral treatment according to the treatment guidelines.
12. Active infections requiring antibiotic intravenous therapy within 1 weeks prior to enrollment.
13. Patients with any other medical conditions that, in the opinion of the Investigator, could affect the patient's participation in the study such as:

    * Disease management may be jeopardized by treatment with this study treatment.
    * Moderate or severe hepatic impairment, i.e., Child-Pugh class B or C.
14. Those who received blood transfusion, albumin, recombinant human thrombopoietin, or colony-stimulating factor therapy within 2 weeks prior to screening.
15. Patients who have not sufficient baseline organ function and whose laboratory data meet the following criteria at enrollment:

    * Absolute Neutrophil Count (ANC) < 1.5×109/L.
    * Total bilirubin > 1.5×ULN.
    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3×ULN without liver metastases or primary liver cancer. AST or ALT > 5×ULN if the patient has documented primary liver cancer or liver metastases.
    * Hemoglobin < 90 g/L.
    * Platelets < 100×109 /L.
    * Creatinine > 1.5×ULN or creatinine clearance < 50 mL/min.
16. Those who are known to be allergic to the active ingredient or excipients of the investigational product BL0020, or who have a predisposition to allergy.
17. Patients with a history of an anaphylactic reaction to irinotecan, irinotecan liposome, or ≥ Grade 3 gastrointestinal toxicity to prior irinotecan, irinotecan liposome.
18. Use of UGT1A1 inhibitors or inducers within 5 half-lives at the time of investigational product BL0020 administration, or planned use of UGT1A1 inhibitors or inducers within 2 weeks prior to administration of BL0020 (whichever is longer), or are expected to continue such therapy during the study.
19. Anti-tumor therapy within 5 half-lives at the time of investigational product BL0020 administration, or anti-tumor therapy within 4 weeks prior to administration of BL0020 (whichever is shorter), therapy including chemotherapy, biologic therapy, immunotherapy, radiotherapy (except palliative radiotherapy and the radiotherapy area do not include the proposed target lesion) and so on, or all relevant toxic reactions (except alopecia) have not been recovered.
20. Patients who are taking anticoagulant therapy (prophylactic use of low-dose aspirin [≤ 100 mg/day] or low molecular weight heparin is allowed).
21. Those who are expected to require systemic corticosteroids within 4 weeks prior to administration of BL0020 (low doses of corticosteroids are excluded, such as ≤ 20 mg prednisone daily or equivalent).
22. Those who have received live or attenuated vaccines (e.g., measles, mumps, rubella, varicella, yellow fever, rabies, BCG, typhoid vaccine, etc.) within 4 weeks before enrollment or scheduled to receive during the study.
23. Those who underwent major surgery within 4 weeks before enrollment, or plan to undergo major surgery during the study.
24. Those who received other investigational drugs within 4 weeks or 5 half-lives of the investigational drugs (whichever is shorter) prior to enrollment.
25. Pregnant or lactating women.
26. Patients who are judged disqualified to join clinical studies by investigator due to any causes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose(MTD) | Throughout the study for approximately 2 years
  Based on the incidence of Dose-Limiting Toxicity (DLT) of BL0020 in patients with advanced solid tumors, MTD is determined.
Recommended Phase II Dose(RP2D) | Throughout the study for approximately 2 years
  RP2D will be evaluated according to all the available safety, PK and efficacy data.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | Cycle 1 day 1 to Cycle 2 day 8
  Area under the plasma concentration time curve
Half life (t1/2) | Cycle 1 day 1 to Cycle 2 day 8
  The elimination half-life time
Disease Control Rate(DCR) | Throughout the study for approximately 2 years
  DCR is defined as the proportion of subjects who achieve a Complete Response (CR) 、Partial Response (PR) or Stable Disease (SD) as assessed by RECIST v1.1
Progression-Free Survival (PFS) | Throughout the study for approximately 2 years
  PFS was defined as the the time from the start date of study treatment to the first documented disease progression or death due to any cause, whichever occurs first.
Duration of overall response (DOR) | Throughout the study for approximately 2 years
  DOR is defined as the time from the first documented CR or PR per RECIST v1.1 to disease recurrence or disease progression (PD) whichever occurs first.
Objective response rate(ORR) | Throughout the study for approximately 2 years
  ORR is defined as the proportion of patients with the best responses of Complete Response (CR) and Partial Response (PR) observed after study treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (3):
  - Cancer Care Foundation Limited, Sydney, New South Wales
  - Scientia Clinical Research, Sydney, New South Wales
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China